CLINICAL TRIAL: NCT05259046
Title: Novel Health Effects of Vitamin K: a Placebo-controlled Randomized Trial in the General Population (InterVitaminK)
Brief Title: The InterVitaminK Trial - Effects of Vitamin K Supplementation on Cardiovascular, Metabolic, and Bone Health
Acronym: InterVitaminK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Director, Professor, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: InterVitaminK
Record Dates: First submitted 2022-01-07; First posted 2022-02-28 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Calcification; Arterial Stiffness
MeSH Terms: interventions — menaquinone 7; Tablets

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a double-blinded manner 1:1 to MK-7 tablets or placebo tablets. Randomisation is conducted in blocks of 6 using computer generated random numbers. A total of 450 participants will be enrolled (225 in each group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, data collectors, and investigators are blinded of the allocation throughout the study period. The randomization list is generated and kept by a statistician employed at the Center for Clinical Research and Prevention, but not involved in the trial. Kappa Bioscience AS, Oslo, Norway, keeps the randomization list for labelling of investigational products. The randomization list will be made available to one DSMB member if safety concerns arise during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention treatment . Dietary supplementation with Menaquinone-7 (MK-7) tablet (333 µg/day). MK-7 (K2VITAL®DELTA) tablets are manufactured by Kappa Bioscience AS, Oslo, Norway.
  Interventions: Dietary Supplement: Menaquinone-7 (MK-7) tablet (333 µg)
- Placebo (Placebo Comparator): Placebo tablet (no active treatment). The placebo tablets will match the intervention treatment in both taste and appearance. Placebo tablets are manufactured by Kappa Bioscience AS, Oslo, Norway.
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Menaquinone-7 (MK-7) tablet (333 µg) — One MK-7 tablet containing 333 µg MK-7 per day
  Arms: Intervention
Dietary Supplement: Placebo tablet — One placebo tablet per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of menaquinone-7 (MK-7) supplementation on cardiovascular, metabolic, and bone health.

DETAILED DESCRIPTION:
Background: Research suggest that vitamin K may have protective effects against non-communicable and age-related diseases as diverse as cardiovascular disease (CVD), osteoporosis, and type 2 diabetes (T2D). However, there is a need for larger studies investigating the potential health effects of vitamin K in the general population.

Objective: The objective of the InterVitaminK trial is to investigate the effects of vitamin K (menaquinone-7, MK-7) supplementation on cardiovascular, metabolic, and bone health.

Hypothesis: The primary hypothesis is that vitamin K supplementation will reduce the progression of coronary artery calcification (CAC) with 15% compared with placebo.

Methods: The InterVitaminK trial is a double-blinded, placebo-controlled, randomized intervention trial. The trial will be conducted in Denmark at the Center for Clinical Research and Prevention and the CT scans will be performed at Rigshospitalet, Denmark. Participants from the Inter99 cohort with detectable CAC (Agatson score >=10) are eligible for the trial. Participants will be randomized 1:1 to receive one daily tablet with MK-7 or placebo for a period of 3 years. Randomization is done in blocks of 6 using computer generated random numbers. Participants are invited for a health examination at baseline and after 1, 2, and 3 years intervention. CT scans are performed at baseline and at 3-year follow-up.

Outcomes: The primary study outcome is progression of CAC from baseline to 3-year follow-up, assessed by Cardiac CT scans. Secondary outcomes are bone mineral density, pulmonary function, and biomarkers of insulin resistance.

Power: Power calculation and sample size considerations are based on the primary endpoint (three-year progression in CAC). A total of 450 participants will be enrolled in the trial. Based on a previous vitamin K trial and data from the Danish cohort study DANCAVAS, it is assumed that the geometric mean three-year progression in CAC in the control group participants is 3.0 with an SD of 1.3. The hypothesis is that vitamin K supplementation can reduce the three-year progression in CAC by 15%. With an estimated dropout-rate of 25% during the study period, a total of 450 participants (225 participants in each group) enrolled at baseline, will provide 89% power to demonstrate an effect of at least 15% (alpha 0.05).

Statistical analyses: The effect of vitamin K supplementation on the primary outcome (CAC) will be analyzed using mixed effects linear regression. The mixed effects linear regression will include a fixed effect for group allocation (intervention/control), a fixed effect for time point (baseline and 3-year follow-up), fixed effect for baseline CAC score and an interaction between group allocation and time point. As baseline measurements are conducted prior to enrolment, treatment at baseline will be modelled as a common treatment category, constraining baseline measurements to no systematic treatment effect between the two arms. The mixed effects model will include a random intercept for each enrolled participant and a first order autoregressive correlation structure allowing correction of measurement for the same participant with higher correlation for measurements closer in time.

Likewise, secondary outcomes and supportive outcomes will be analyzed using mixed effects linear regression. Analysis and presentation of data will be in accordance with the CONSORT guidelines. For details, see the statistical analysis plan uploaded at clinicaltrials.gov (NCT05259046).

ELIGIBILITY:
Inclusion Criteria:

* Detectable CAC (Agatson score >=10) assessed by Cardiac Computed Tomography (CT) scan in the Inter99 20-year follow-up study

Exclusion Criteria:

* Manifest CVD (prior cerebral infarct, prior myocardial infarct, prior percutaneous coronary intervention or prior coronary artery bypass surgery)
* Noise on the CT scan, which complicates an accurate assessment of CAC and interpretation of the CT scan. An example is a pacemaker
* Current treatment with Vitamin K antagonist (VKA).
* History of coagulation disorders (hemophilia, von Willebrand disease, sickle cell anemia)
* Active malignant disease (ongoing treatment)
* Previous surgical removal of the thyroid gland, or one or more of the parathyroid glands
* Regular use of vitamin K supplements other than trial tablets
* Pregnancy or breastfeeding

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Total coronary artery calcification | Baseline to three years of follow-up
  Total coronary artery calcification score (unit: Agatston score) in the coronary arteries, assessed by non-contrast Cardiac CT scans. A high score reflects higher degree of calcification in the coronary arteries and increased risk of coronary artery disease. The outcome will be evaluated by randomization group (active versus placebo).

SECONDARY OUTCOMES:
Coronary plaque composition | Baseline to three years of follow-up
  Total coronary plaque composition (calcified, non-calcified subcomponents) assessed by contrast Cardiac CT scans (unit: cubic millimeters)
Arterial stiffness | Baseline to three years of follow-up
  Arterial stiffness assessed by carotid-femoral pulse wave velocity examination (unit: meters/second)
Blood pressure | Baseline to three years of follow-up
  Blood pressure (unit: millimeter of mercury) assessed by a digital blood pressure device. Both systolic and diastolic blood pressure will be evaluated.
Aortic valve calcifications | Baseline to three years of follow-up
  Aortic valve calcifications assessed by non-contrast Cardiac CT scans (unit: Agatston score). A high score reflects higher degree of calcification
Bone mineral density | Baseline to three years of follow-up
  Bone mineral density assessed by quantitative CT scan of the columna thoracalis (unit: milligrams/cubic centimeter)
Pulmonary function | Baseline to three years of follow-up
  Pulmonary function reflected by forced expiratory volume in one second (FEV1) (unit: Volume in Liter)
Insulin resistance | Baseline to three years of follow-up
  Insulin resistance assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) (unit: millimoles/liter * picomoles/liter)

OTHER OUTCOMES:
Biomarkers of bone resorption | Baseline to three years of follow-up
  Bone metabolism reflected by biomarkers of bone resorption including C-terminal telopeptide of type I collagen (CTX) (unit: picograms/milliliter)
Biomarkers of bone formation | Baseline to three years of follow-up
  Bone metabolism reflected by biomarkers of bone formation including osteocalcin (with different phosphorylation and carboxylation forms) (unit: nanograms/milliliter), Fibroblast growth factor 23 (FGF23) (unit: nanograms/milliliter), osteoprotegerin (unit: Picomoles/liter), and Procollagen 1 Intact N-Terminal Propeptide (P1NP) (unit: milligram/liter)
Lung function | Baseline to three years of follow-up
  Lung function reflected by expiratory forced vital capacity (FVC) and FEV1/FVC-ratio
Lung tissue density | Baseline to three years of follow-up
  Lung tissue density as a measure of lung fibrosis assessed by CT scan
Respiratory infections | Baseline to three years of follow-up
  Annual number of respiratory infectious disease episodes, both upper and lower respiratory infections including COVID-19 (registered through telephone interviews)
Glucose control | Baseline to three years of follow-up
  Glucose metabolism reflected by Glycated hemoglobin A1c (HbA1c) (unit: millimole/mol)
Lipid metabolism | Baseline to three years of follow-up
  Lipid metabolism biomarkers (including total cholesterol, triglycerides, low-density lipoprotein, high-density lipoprotein) (unit: milligrams/deciliter)
Inflammation | Baseline to three years of follow-up
  Inflammatory biomarkers including interleukin-6 (IL-6) (unit: picograms/milliliter) and Tumor necrosis factor α (TNF-α) (unit: picograms/milliliter).
Body composition | Baseline to three years of follow-up
  Anthropometry reflected by body fat percentage (%) assessed by bioimpedance (unit is estimated per cent fat mass).

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Research and Prevention, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No
After the publication of the main results upon completion of the trial, data will be available on a collaborative basis following approval from the InterVitaminK Trial Steering Committee and the regional data protection authority.

REFERENCES:
- [Derived] Kampmann FB, Thysen SM, Nielsen CFB, Kofoed KF, Kober L, Pham MHC, Vaag A, Jorgensen NR, Petersen J, Jacobsen RK, Karhus LL, Diederichsen A, Frimodt-Moller M, Linneberg A. Study protocol of the InterVitaminK trial: a Danish population-based randomised double-blinded placebo-controlled trial of the effects of vitamin K (menaquinone-7) supplementation on cardiovascular, metabolic and bone health. BMJ Open. 2023 May 19;13(5):e071885. doi: 10.1136/bmjopen-2023-071885. PMID 37208133

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT05259046/SAP_000.pdf